CLINICAL TRIAL: NCT06724016
Title: A Phase I, Open-Label, Multicenter, Dose Escalation and Expansion Study of HM16390, as a Single Agent and in Combination With Pembrolizumab, in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Dose Escalation and Expansion Study of HM16390 Alone or With Pembrolizumab in Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM-LIL2-101; KEYNOTE-G39 (Other: Merck & Sharp Dohme LLC); MK-3475-G39 (Other: Merck & Sharp Dohme LLC)
Record Dates: First submitted 2024-11-29; First posted 2024-12-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: 1. Dose-Escalation Part: Divided into 2 arms (Arm A: HM16390 monotherapy, Arm B: HM16390 in combination with pembrolizumab)
  2. Dose-Ranging Part: Subjects will be randomized 1:1 into at least two dose levels to enable better selection of the doses for further evaluation, and may apply to cohorts of both monotherapy and combination therapy
  3. Dose-Expansion Part: Based on the available data from Dose-Escalation and Dose-Ranging parts, the most feasible dose will be selected as the RDE and will be administered to subjects in indication-specific expansion cohorts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HM16390 (Experimental): HM16390 Monotherapy
  Interventions: Drug: HM16390
- HM16390 + pembrolizumab (Experimental): HM16390 in combination with pembrolizumab
  Interventions: Drug: HM16390; Drug: pembrolizumab

INTERVENTIONS:
Drug: HM16390 — HM16390 will be administered subcutaneously using syringes on Day 1 of every 3-week treatment cycle
Drug: pembrolizumab — Fixed dose of pembrolizumab will be administered as an IV infusion over 30 minutes on Day 1 of every 3-week treatment cycle
  Other Names: KEYTRUDA®
  Arms: HM16390 + pembrolizumab

SUMMARY:
This is a First-in-Human, Phase 1, Dose-Escalation and Dose-Expansion study of HM16390, as a single agent and in combination with pembrolizumab to assess safety, tolerability, MTD, RP2D, PK, and efficacy in patients with advanced or metastatic solid tumors.

Dose-Escalation Part is planned to establish the MTD or RDs for the randomized Dose-Ranging Part. Based on the results of the Dose-Escalation Part, additional eligible subjects will be randomized 1:1 into each dose level. After a comprehensive review of available data from both Dose-Escalation Part and Dose-Ranging Part, the RDEs to be tested in the Dose-Expansion Part are determined. Dose-Expansion Part is designed to assess the potential efficacy of HM16390 as a single agent and in combination with pembrolizumab when administered at the RDEs to subjects in indication-specific expansion cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a histologically and/or cytologically confirmed advanced or metastatic solid tumor and have failed or are intolerant to standard therapy with clinical benefit.
* Patients in the Dose-Escalation Part must have evaluable or measurable disease at baseline and the patients for Dose-Ranging and Dose-Expansion Part must have at least one measurable lesion at baseline by computed tomography (CT) or magnetic resonance imaging (MRI) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 assessed within 7 days before allocation or randomization.
* Age of 18 years or older (or country's legal age of majority if the legal age was >18 years)
* Adequate renal function.
* Adequate hematologic function.
* Adequate liver function.

Key Exclusion Criteria:

* Received prior treatment with agent targeting the IL-2, IL-7, or IL-15 receptors, or related to mode of action of HM16390.
* Known active CNS metastases and/or carcinomatous meningitis.
* History of severe toxicities associated with a prior immunotherapy.
* Any prior treatment-related (i.e. chemotherapy, immunotherapy, radiotherapy) clinically significant toxicities that have not resolved to Grade ≤ 1 per NCI-CTCAE version 5.0 or prior treatment-related toxicities that are clinically unstable and clinically significant at time of enrollment.
* Has ongoing or suspected autoimmune disease.
* Known active and clinically significant bacterial, fungal or viral infection including known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, immunocompromised patients.
* History of chronic liver disease or evidence of hepatic cirrhosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2031-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Incidence and nature of DLTs | At the end of Cycle 1 (each cycle is 21 days) in Dose-Escalation Part
  To evaluate safety and tolerability of HM16390 as a single agent and in combination with pembrolizumab
Incidence, nature, and severity of adverse events and laboratory abnormalities graded per NCI-CTCAE v5.0. | Throughout the study until end of safety follow-up period (90 days after the last treatment)
  To evaluate safety and tolerability of HM16390 as a single agent, and in combination with pembrolizumab

SECONDARY OUTCOMES:
The maximum serum concentration (Cmax) | Throughout the study until treatment discontinuation (up to 2-3 years)
  To evaluate PK profile upon HM16390 administration
The time to reach Cmax (Tmax) | Throughout the study until treatment discontinuation (up to 2-3 years)
  To evaluate PK profile upon HM16390 administration
The area under the concentration-time curve from time 0 to the last observable concentration (AUClast) | Throughout the study until treatment discontinuation (up to 2-3 years)
  To evaluate PK profile upon HM16390 administration
The AUC extrapolated to infinity (AUCinf) | Throughout the study until treatment discontinuation (up to 2-3 years)
  To evaluate PK profile upon HM16390 administration
The AUC during the dosing interval (AUCtau) | Throughout the study until treatment discontinuation (up to 2-3 years)
  To evaluate PK profile upon HM16390 administration
The serum concentration at the end of the dosing interval (Ctrough) | Throughout the study until treatment discontinuation (up to 2-3 years)
  To evaluate PK profile upon HM16390 administration
The elimination half-life (T1/2) | Throughout the study until treatment discontinuation (up to 2-3 years)
  To evaluate PK profile upon HM16390 administration
The apparent volume of distribution (Vd/F) | Throughout the study until treatment discontinuation (up to 2-3 years)
  To evaluate PK profile upon HM16390 administration
The apparent clearance (CL/F) | Throughout the study until treatment discontinuation (up to 2-3 years)
  To evaluate PK profile upon HM16390 administration
Objective response rate (ORR) | Throughout the study until disease progression or death whichever occurs first (up to 2-3 years)
  ORR will be measured as the proportion of subjects with a confirmed response of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Disease Control Rate (DCR) | Throughout the study until disease progression or death whichever occurs first (up to 2-3 years)
  DCR will be measured as the proportion of subject with confirmed CR, PR, or Stable Disease (SD) as per RECIST v1.1
Progression-free survival (PFS) | Throughout the study until disease progression or death whichever occurs first (up to 2-3 years)
  PFS will be measured from date of first treatment until date of radiographic progression as per RECIST v1.1 or until death from any cause, whichever occurs first
Duration of response (DOR) | Throughout the study until disease progression or death whichever occurs first (up to 2-3 years)
  DOR will be measured as the time from initial onset of CR or PR to first radiographic progression as per RECIST v1.1 or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No